CLINICAL TRIAL: NCT01777815
Title: Safety and Performance Study of the NeoChord Suturing Device in Subjects With Degenerative Mitral Valve Disease; Diagnosed With Severe Mitral Regurgitation
Brief Title: Safety and Performance Study of the NeoChord Device
Acronym: TACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoChord (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-610404-100; 09/1819 (Other: FEKI)
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Mitral Valve Regurgitation
Keywords: NeoChord; DS1000; Mitral Valve; Mitral Valve Regurgitation; MR; Mitral Valve Repair; Mitral Valve Prolapse; Artificial Chordae
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implanting ePTFE sutures (Experimental): Implanting ePTFE sutures as artificial neochordae using the NeoChord DS1000 Artificial Chordae Delivery System
  Interventions: Device: NeoChord DS1000 Artificial Chordae Delivery System

INTERVENTIONS:
Device: NeoChord DS1000 Artificial Chordae Delivery System

SUMMARY:
The purpose of this study is to demonstrate the safety and performance of the NeoChord DS1000 Artificial Chordae Delivery System in implanting ePTFE sutures(s) as artificial neochordae in patients with mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 and < 80 years
* Candidate for surgical mitral valve repair or replacement
* Isolated posterior leaflet prolapse
* Moderate to severe or severe mitral valve regurgitation that is degenerative in nature

Exclusion Criteria:

* Anterior or bi-leaflet prolapse
* Functional or ischemic MR
* NYHA Class IV
* Complex mechanism of MR (leaflet perforation, etc)
* Significant tethering of leaflets toward LV apex
* Severely calcified mitral valve annulus
* Inflammatory valve disease
* Severe LV dilation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Procedural Success | 30 days
  The placement of at least one neochord using the DS1000 System AND a reduction in mitral regurgitation <= 2+ at the time of the procedure AND maintained MR reduction of <= 2+ at 30 days

SECONDARY OUTCOMES:
Procedural Safety | 30 days
  the rate of Major Adverse Events (MAE) defined as a combined endpoint of: death, MI, reoperation for failed surgical repair, non-elective cardiovascular surgery to treat an adverse event, procedural ventilation > 48 hours, procedure-related transfusion of > 2 units blood product, stroke, renal failure, deep wound infection, new onset of permanent AF, and septicemia, through 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Anno Diegeler, MD, Principal Investigator — Herz und Gefäß-Klinik
Locations (8):
- Aarhus University Hospital, Skejby, Aarhus, Denmark
- Germany (4):
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz und Gefäß-Klinik, Bad Neustadt an der Saale
  - Herzzentrum Leipzig, Leipzig
  - Klinik für Herz-und Gefäßchirurgie, Munich
- Italy (2):
  - San Raffaele, Milan
  - Ospedale San Giovanni Battista "Molinette", Torino
- Vilniaus Universiteto ligonines Santariskiu, Vilnius, Lithuania

REFERENCES:
- [Derived] Seeburger J, Rinaldi M, Nielsen SL, Salizzoni S, Lange R, Schoenburg M, Alfieri O, Borger MA, Mohr FW, Aidietis A. Off-pump transapical implantation of artificial neo-chordae to correct mitral regurgitation: the TACT Trial (Transapical Artificial Chordae Tendinae) proof of concept. J Am Coll Cardiol. 2014 Mar 11;63(9):914-9. doi: 10.1016/j.jacc.2013.07.090. Epub 2013 Sep 24. PMID 24076529